CLINICAL TRIAL: NCT07002957
Title: Spiritual Music Therapy for Individuals on Probation: A Mixed-Method Randomised Controlled Trial
Brief Title: Spiritual Music Therapy for Individuals on Probation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Gonca Ustun, Associate Professor, Amasya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Spiritual Music Therapy
Record Dates: First submitted 2025-05-01; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Music Therapy; Spirituality; Prisoners
Keywords: Music Therapy; Spirituality; Probation

STUDY DESIGN:
Intervention Model Description: Mixed methods randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In the study, the intervention group received six 90-minute sessions of spiritual music therapy once a week. The groups consisted of 14 participants and the study was completed in five groups.
  Interventions: Other: Spiritual Music Therapy
- Control group (No Intervention): No intervention was made to the control group.

INTERVENTIONS:
Other: Spiritual Music Therapy — In the first session of the spiritual music therapy application, information was given about music, music therapy and its history, and information was given about the Turkish Music makam structure and makam differences and the traces these makams leave on the person's body and soul. In addition, the technique of receiving and giving sound was taught. In the next five sessions, Rast, Uşşak, Segâh, Hüseyni and Hicaz makams were listened to, accompanied by the sound of kanun and water. Information was given about the musical and therapeutic status of the makams, 3 works related to the relevant makam were taught, performed and information was given about the spiritual messages of the piece, its composer and lyricist. At the same time, rhythm studies were done with the bendir to accompany the relevant makam. At the end of each session, the makam of the day was listened to, accompanied by the sound of kanun and water.
  Arms: Intervention group

SUMMARY:
The purpose of this research is to determine the effect of spiritual music therapy application on the state and trait anxiety, self-esteem and depression levels of individuals on probation and to evaluate the effectiveness of spiritual music therapy application.

The basic questions of the study are as follows; What did the spiritual music therapy application make you feel? Did it have an effect on state and trait anxiety, self-esteem and depression? The intervention group received 6 weeks of spiritual music therapy by the researcher. Data were collected before and after the intervention. The effect of the intervention was evaluated with open-ended questions. The control group was not treated.

DETAILED DESCRIPTION:
In this mixed-method randomized controlled study, individuals on probation who were tried for the same crime were randomly assigned to the intervention (spiritual music therapy) group and the control group in a 1:1 ratio. The study was approved by the Amasya University Non-Interventional Clinical Research Ethics Committee (decision numbered 2024/84) and the Amasya Probation Office (decision numbered 2024/926). The study was prepared in accordance with the CONSORT 2010 guide. The study sample consisted of 140 participants who were subject to probation in accordance with Article 191 of the Turkish Penal Code (Purchasing, accepting or possessing drugs or stimulants for use or using drugs or stimulants) at the Amasya Probation Office between April 2024 and March 2025. In the study, which included individuals over the age of 18, participants whose probation period ended (file closed), who went to prison or who changed their address were excluded from the study. The study was completed with 46 participants in the intervention group and 45 participants in the control group. In the study, six 90-minute sessions of spiritual music therapy were applied to the intervention group once a week. The groups consisted of 14 participants and the study was completed in five groups. No intervention was made to the control group, the group only came for control purposes. The spiritual music therapy application was carried out by the researcher. The applications were carried out in a circular seating plan in an education hall with a fountain in the middle. During the sessions, water sounds, kanun, bendir and musical notes were used. In the first session, information was given about music, music therapy and its history, and information was given about the Turkish Music makam structure and makam differences and the traces these makams leave on the person's body and soul. In addition, the technique of receiving and giving sound was taught. In the next five sessions, Rast, Uşşak, Segâh, Hüseyni and Hicaz makams were listened to with the sound of kanun and water, respectively. Information was provided about the musical and therapeutic status of the modes, 3 pieces related to the relevant mode were taught, performed and information was provided about the spiritual messages, composer and lyricist of the piece. At the same time, rhythm studies were performed with the bendir to accompany the relevant mode. At the end of each session, the mode of the day was listened to with the sound of kanun and water. The primary outcome measurements of the study were made weekly and evaluated at the end of each session. The secondary outcome measurements were completed at the end of each six-week application. The application area, the researcher who carried out the application, the application methods, the researcher who carried out the data collection process and the groups of the participants did not change for any reason and the same protocol was applied until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Implementation of probation pursuant to Article 191 of the Turkish Penal Code (Purchasing, accepting or possessing narcotic or stimulant substances for use or using narcotic or stimulant substances)

Exclusion Criteria:

* those whose probation period has ended (whose file has been closed)
* those who have entered prison
* those who have changed their address

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
End-of-session qualitative assessment | During the intervention
  Spiritual music therapy was applied to 5 groups of 14 participants once a week for 6 sessions. At the end of each session, the effect of the theme covered that week on the participants was measured by asking a structured questionnaire consisting of 2 questions. These questions were; How did the theme covered in this session make you feel? What feelings and thoughts did this session evoke in you? The data was evaluated qualitatively. analyzed. As the primary outcome measure, it was expected that the participants would experience positive feelings at the end of the weekly application.
State and Trait Anxiety Inventory- Pre test | At the time of enrollment
  Developed by Spielberger et al. (1970), it was adapted to Turkish by Öner and Le Compte (1985). State Anxiety Inventory (STAI-1) reveals how a person feels at a certain moment and under certain conditions. Trait Anxiety Inventory (STAI-2) determines how an individual feels, independent of the environment and conditions they are in. There are 40 propositions that individuals can use to express their feelings in the State and Trait Anxiety Inventory. Depending on how the person feels and the severity of their feelings, they should mark one of the following options: "Not at all" (1), "A little" (2), "A fair amount" (3), "Completely" (4). A high score indicates a high level of anxiety, while a low score indicates a low level of anxiety. Cronbach's Alpha values of the scale were determined as 0.83-0.92 for the state anxiety scale and 0.83-0.87 for the trait anxiety scale. It was measured before treatment for both the intervention and control groups.
Rosenberg Self-Esteem Scale -Pre test | At the time of enrollment
  Developed by Rosenberg (1965), its Turkish validity and reliability were made by Çuhadaroğlu (1986). The scale is a self-report scale consisting of 63 questions. The scale consists of 12 subcategories. The first 10 items of the scale are used to measure self-esteem. Five of these items are positive and five are negative. It is a Likert-type scale consisting of the options "Very True", "True", "False" and "Very False". According to the evaluation system within the scale; questions 1, 2, 4, 6, 7 are positive and scored from 3 to 0, while questions 3, 5, 8, 9, 10 are negative and scored from 0 to 3. The total score range is between 0-30 points, and a score below 15 points indicates low self-esteem. The Cronbach's Alpha value of the scale is 0.75. It was measured before treatment for both the intervention and control groups.
Beck Depression Inventory -Pre test | At the time of enrollment
  The scale developed by Beck and colleagues (1961) is a self-assessment scale consisting of 21 questions used to measure depressive symptoms in areas such as cognitive and emotional coping skills. Each item of the scale aims to measure the degree of symptoms specific to depression, and each item contains self-assessment sentences scored between 0-3 on a four-point Likert type that can describe depressive symptoms in the last week. The total score range on the scale varies between 0-63. The Turkish adaptation was made by Hisli (1989). The Cronbach's Alpha value of the scale was found to be 0.80. It was measured before treatment for both the intervention and control groups.

SECONDARY OUTCOMES:
Qualitative evaluation after intervention | At the end of the 6-week treatment
  Spiritual music therapy was applied to 5 groups of 14 participants once a week for 6 sessions. After all the sessions were completed, a face-to-face interview was conducted with the participants about how this application made them feel; how it affected their emotions, thoughts and behaviors, relationships and harmony within the group; and semi-structured questions that allowed them to express the most impressive and most negative aspects of the application. As the secondary outcome measure, it was expected that the participants would experience positive emotions at the end of the weekly application.
State-Trait Anxiety Scale-Post test | At the end of the 6-week treatment
  After all the sessions were completed the State-Trait Anxiety Scale was conducted with the participants. Developed by Spielberger et al. (1970), it was adapted to Turkish by Öner and Le Compte (1985). State Anxiety Inventory (STAI-1) reveals how a person feels at a certain moment and under certain conditions. Trait Anxiety Inventory (STAI-2) determines how an individual feels, independent of the environment and conditions they are in. There are 40 propositions that individuals can use to express their feelings in the State and Trait Anxiety Inventory. Depending on how the person feels and the severity of their feelings, they should mark one of the following options: "Not at all" (1), "A little" (2), "A fair amount" (3), "Completely" (4). A high score indicates a high level of anxiety, while a low score indicates a low level of anxiety. Cronbach's Alpha values of the scale were determined as 0.83-0.92 for the state anxiety scale and 0.83-0.87 for the trait anxiety scale.
Rosenberg Self-Esteem Scale -Post test | At the end of the 6-week treatment
  After all the sessions were completed the Rosenberg Self-Esteem Scale was conducted with the participants. Developed by Rosenberg (1965), its Turkish validity and reliability were made by Çuhadaroğlu (1986). The scale is a self-report scale consisting of 63 questions. The scale consists of 12 subcategories. The first 10 items of the scale are used to measure self-esteem. Five of these items are positive and five are negative. It is a Likert-type scale consisting of the options "Very True", "True", "False" and "Very False". According to the evaluation system within the scale; questions 1, 2, 4, 6, 7 are positive and scored from 3 to 0, while questions 3, 5, 8, 9, 10 are negative and scored from 0 to 3. The total score range is between 0-30 points, and a score below 15 points indicates low self-esteem. The Cronbach's Alpha value of the scale is 0.75.
Beck Depression Inventory -Post test | At the end of the 6-week treatment
  After all the sessions were completed the Beck Depression Inventory was conducted with the participants. Beck Depression Inventory: The scale developed by Beck and colleagues (1961) is a self-assessment scale consisting of 21 questions used to measure depressive symptoms in areas such as cognitive and emotional coping skills. Each item of the scale aims to measure the degree of symptoms specific to depression, and each item contains self-assessment sentences scored between 0-3 on a four-point Likert type that can describe depressive symptoms in the last week. The total score range on the scale varies between 0-63. The Turkish adaptation was made by Hisli (1989). The Cronbach's Alpha value of the scale was found to be 0.80.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No